CLINICAL TRIAL: NCT05076708
Title: The Effects of IQOS Use on Cigarette Smoking Behaviors
Acronym: IQOS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Janet Audrain-McGovern, Professor, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 843646
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Smoking; Cigarette Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Cigarette Smoking; Tobacco Use

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IQOS (Other)
  Interventions: Other: IQOS

INTERVENTIONS:
Other: IQOS — All participants switch from cigarette smoking to IQOS use for a 14-day phase.

SUMMARY:
This within-subjects study aims to evaluate the effects of IQOS use on combustible cigarette smoking behaviors among 100 cigarette smokers who completed the study. After measuring baseline cigarette smoking rate, participants will receive an IQOS device and be instructed to use it (versus cigarettes) over a 14-day period. The investigators will also examine which objective and subjective effects of IQOS use predict a complete and incomplete switch from cigarettes to IQOS.

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate fluently in English (i.e. speaking, writing, and reading).
2. Male and female smokers who are between 18 and 65 years of age and self-report smoking at least 5 cigarettes (menthol and/or non-menthol) per day for at least the last 12 months.
3. Not currently undergoing smoking cessation treatment or planning to quit smoking within the next 30 days.
4. Report an interest in quitting smoking within the next 6 months.
5. Plan to live in the area for the duration of the study
6. Willing to use study provided IQOS devices and HeatSticks during 2 laboratory visits and throughout study participation.
7. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.

Exclusion Criteria:

Smoking Behavior

1. Regular use of nicotine containing products other than cigarettes (e.g. chewing tobacco, snuff, snus, cigars, e-cigs, etc.). Participants agreeing to abstain from using nicotine containing products other than cigarettes for the duration of study will be considered eligible.
2. Current enrollment or plans to enroll in a smoking cessation program over the duration of the study (i.e. 21 days/3 weeks).
3. Provide a CO breath test reading less than 10 ppm at Intake.

Alcohol and Drug

1. History of substance abuse (other than nicotine dependence) in the past 12 months and/or currently receiving medical treatment for substance abuse. Counseling and support groups (e.g. Alcoholics Anonymous and Narcotics Anonymous) will not be considered medical treatment for the purposes of this protocol.
2. Current alcohol consumption that exceeds 20 standard drinks/week.
3. Breath alcohol reading (BrAC) greater than .000 at Intake.

Medical

1. Women, including all individuals assigned as "female" at birth, who are pregnant, breast feeding, or planning a pregnancy over the duration of the study period.
2. Serious or unstable disease within the past year (e.g. cancer, heart disease). Applicable conditions will be evaluated on a case-by-case basis by the Principal Investigator.

Psychiatric

1. Lifetime history of schizophrenia or psychosis.
2. Lifetime history or current diagnosis of active major depression. Participants who maintain a diagnosis of major depression who have not experienced any major depressive episodes in the past 6 months and are stable on antidepressant medication(s) are eligible to participate.
3. Lifetime history of a suicide attempt.

General Exclusion

1. Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact subject safety, study data, and/or the study design as determined by the Principal Investigator.
2. Any medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator. Subjects may be deemed ineligible for any of the aforementioned reasons at any point throughout the study, as well as during the initial telephone screen.
3. Significant non-compliance with protocol and/or study design as determined by the Principal Investigator and/o. Subjects may be deemed ineligible at any point throughout the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Audrain-McGovern J, Wileyto EP, Klapec O, Koita F, Strasser AA. Switching from cigarettes to IQOS: the relative importance of IQOS-associated reward, reinforcement and abstinence relief. Tob Control. 2025 Oct 3;34(5):651-658. doi: 10.1136/tc-2024-058635. PMID 38871445

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IQOS
Started | 102
Completed | 90
Not Completed | 12
Not completed — Withdrawal by Subject | 4
Not completed — Lost to study during switch phase | 8

BASELINE CHARACTERISTICS:
Arm/Group | IQOS
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.20 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 53
  White | 32
  Other | 5
Baseline Smoking Rate [Mean (Standard Deviation); unit: cigarettes per day] — Participants eligible at the intake screening completed baseline measures and received instructions to smoke as usual for the next 5 days while collecting all spent filters each day (days 1-5). The average daily spent filters served as the baseline smoking rate.
  cigarettes per day | 13.40 (6.06)
Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Nicotine dependence was measured using The Fagerstrom Test for Nicotine Dependence (FTND). The FTND is a 6-item scale with higher scores indicating greater levels of nicotine dependence. Nicotine dependence scores can range from 0 (low) to 8 (high).
  units on a scale | 5.11 (1.91)
Subjective Reward [Mean (Standard Deviation); unit: units on a scale] — The subjective rewarding value of IQOS was measured by averaging the two-item satisfaction subscale ('Was it satisfying'? and 'Did it taste good'?) from the Cigarette Evaluation Scale (CES) adapted for IQOS use. The CES is an 11 item Likert-format (1=not at all to 7=extremely) self-report instrument. The minimum possible score is 2 and the maximum is 14. Higher scores denote greater subjective rewarding value.
  units on a scale | 8.01 (3.16)
Relative Reinforcing Value [Mean (Standard Deviation); unit: trials] — Using a validated computer choice task, participants chose between clicking one image to earn points for IQOS puffs (25 clicks to earn a point for a puff) or another image to earn points for cigarette puffs (25x clicks to earn a point for a puff) across 10 trials. The breakpoint, the highest trial (range 0-10) completed to earn cigarette puffs indicates the reinforcing value of cigarettes relative to IQOS. Working for cigarette puffs on <5 trials equate to a lower reinforcing value of cigarettes, whereas working on 5 or more trials reflects higher reinforcing value of cigarettes.
  trials
    Breakpoint | 7.69 (3.21)
    Lower<5 | 1.88 (1.58)
    Higher>5 | 9.04 (1.53)
Withdrawal Symptom Relief [Mean (Standard Deviation); unit: units on a scale] — Participants completed 10-hours of abstinence before trying IQOS. Withdrawal symptoms were measured by summating the 8-item Minnesota Nicotine Withdrawal Scale (MNWS). MNWS Likert response options are 0=none to 4=severe; score range=0-32). Higher scores indicate greater withdrawal symptoms. Withdrawal relief scores were calculated as post-IQOS use minus pre-IQOS use scores. The relief score represents the level of withdrawal symptom relief after IQOS use.
  units on a scale | -1.73 (3.74)
Craving Relief [Mean (Standard Deviation); unit: units on a scale] — Participants completed 10 hours of abstinence before trying IQOS. Craving was measured with the well-validated and reliable 4-item Negative reinforcement subscale of the brief Questionnaire of Smoking Urges (QSU-brief). Likert response options ranged from 1=strongly disagree to 7=strongly agree. Scores were calculated by summating the 4 items (range=4-28). Higher scores indicate greater cigarette cravings. A craving relief score was calculated as post-IQOS use score minus pre-IQOS use score.
  units on a scale | -4.10 (6.11)

OUTCOME MEASURES:

1. Primary Outcome: Cigarette Consumption
Description: The primary outcome was the count of cigarettes per day (CPD) across the 14-day switch period (days 8-21) compared with the average CPD at baseline (days 1-5). This outcome was determined by counting each daily spent cigarette filter returned and self-reported CPD. The correlation between self-report and spent filter return was r=0.98. For the analysis, the daily counts were transformed to a percentage of the participant's average smoking rate from the baseline ad-lib smoking period.
Time Frame: Day 1-Day 21 (21 days)
Measure: Mean (95% Confidence Interval); unit: percentage of baseline smoking rate
Arm/Group | IQOS
Number analyzed (Participants) | 90
percentage of baseline smoking rate | 31.68 [7.82 to 55.54]

2. Secondary Outcome: Change in Motivation to Quit Smoking
Description: Motivation to quit smoking was measured at baseline (day 1) and study end (day 21) using the contemplation ladder (0 = no thoughts of quitting to 10 = taking action to quit). A summary change score was generated by subtracting the baseline measure from the measure at study end.
Time Frame: Day 1-Day 21 (21 days)
Population: The 90-participant sample was reduced to 87, with 3 subjects missing the contemplation ladder measure at the end of the study.
Measure: Mean (Standard Deviation); unit: ladder steps
Arm/Group | IQOS
Number analyzed (Participants) | 87
ladder steps | 1.47 (1.98)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Adverse Events were defined as any unexpected event related to IQOS use.
  Serious Adverse Events were defined as any severe or serious event related to IQOS use.
Arm/Group | IQOS
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT05076708/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT05076708/ICF_001.pdf